CLINICAL TRIAL: NCT03777059
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Safety, and Tolerability of Oral Atogepant for the Prevention of Migraine in Participants With Episodic Migraine (ADVANCE)
Brief Title: 12-Week Placebo-controlled Study of Atogepant for the Preventive Treatment of Migraine in Participants With Episodic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3101-301-002
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Episodic Migraine
Keywords: Migraine; Aura
MeSH Terms: conditions — Migraine Disorders; Epilepsy | interventions — atogepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo-matching atogepant tablets orally once daily for 12 weeks.
  Interventions: Drug: Placebo
- Atogepant 10 mg (Experimental): Atogepant 10 mg tablet orally once daily and placebo-matching atogepant tablets orally once daily for 12 weeks.
  Interventions: Drug: Atogepant; Drug: Placebo
- Atogepant 30 mg (Experimental): Atogepant 30 mg tablet orally once daily and placebo-matching atogepant tablets orally once daily for 12 weeks.
  Interventions: Drug: Atogepant; Drug: Placebo
- Atogepant 60 mg (Experimental): Atogepant 60 mg tablet orally once daily and placebo-matching atogepant tablets orally once daily for 12 weeks.
  Interventions: Drug: Atogepant; Drug: Placebo

INTERVENTIONS:
Drug: Atogepant — Atogepant tablet
  Arms: Atogepant 10 mg; Atogepant 30 mg; Atogepant 60 mg
Drug: Placebo — Placebo-matching atogepant tablets

SUMMARY:
To evaluate the safety and tolerability of atogepant 30 mg and 60 mg once a day for the prevention of migraine in participants with episodic migraine.

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of migraine with or without aura consistent with a diagnosis.
* Age of the participant at the time of migraine onset <50 years.

Exclusion Criteria:

* Has a history of migraine accompanied by diplopia or decreased level of consciousness or retinal migraine.
* Has a current diagnosis of chronic migraine, new persistent daily headache, trigeminal autonomic cephalgia (e.g., cluster headache), or painful cranial neuropathy.
* History of an inadequate response to >4 medications (2 of which have different mechanisms of action) prescribed for the prevention of migraine.
* Participants with clinically significant hematologic, endocrine, cardiovascular, pulmonary, renal, hepatic, gastrointestinal, or neurologic disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 910 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Trugman, MD, Study Director — Allergan
Locations (136):
- United States (136):
  - Synexus Clinical Research US, Inc., Chandler, Arizona
  - Advanced Research Associates, Glendale, Arizona
  - Alea Research Institute, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Orange Grove Family Practice, Tucson, Arizona
  - Principals Research Group, Hot Springs, Arkansas
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Med Center Medical Clinic, Carmichael, California
  - Triwest Research Associates, El Cajon, California
  - Neuro Pain Medical Center, Fresno, California
  - California Headache and Balance Center, Fresno, California
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Neurology Center of North Orange County, Fullerton, California
  - NervePro Research Bruce Cleeremans, Irvine, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - Long Beach Clinical Trials Services, Long Beach, California
  - Keck Medicine of USC, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - Newport Beach Clinical Research Associates, Newport Beach, California
  - Excell Research, Inc., Oceanside, California
  - Stanford, Palo Alto, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - Desert Valley Research, Redlands, California
  - George J. Rederich, M.D. Inc., Redondo Beach, California
  - Paradigm Clinical Research Centers, Inc, San Diego, California
  - Optimus Medical Group, San Francisco, California
  - California Neuroscience Research, Sherman Oaks, California
  - Synexus Clinical Research US, Inc., Vista, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Delta Waves, Inc., Colorado Springs, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Aventura Neurological Associates, Aventura, Florida
  - Neurology Offices of South Florida, Boca Raton, Florida
  - Sarkis Clinical Trials- Gainesville, Gainesville, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Neurology Associates, P.A., Maitland, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Sarasota Memorial Hospital Clinical Research Center, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Neurotrials Research, Atlanta, Georgia
  - Pediatric and Adolescent NeuroDevelopmental Associates (PANDA) Neurology, Atlanta, Georgia
  - Synexus Clinical Research US, Inc., Atlanta, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Diamond Headache Clinic Ltd, Chicago, Illinois
  - Clinical Investigation Specialists, Gurnee, Illinois
  - JWM Neurology, Indianapolis, Indiana
  - Deaconess Clinic - Gateway Health Center, Newburgh, Indiana
  - PMG Research, Inc. d/b/a PMG Research of McFarland Clinic, Ames, Iowa
  - Heartland Research Associates, LLC, Newton, Kansas
  - College Park Family Care Center, Overland Park, Kansas
  - Phoenix Medical Research, Prairie Village, Kansas
  - Heartland Research Associates, LLC - An AMR Company, Wichita, Kansas
  - Ochsner Clinic Foundation, Covington, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Mid-Atlantic Permanente Medical Group, PC, Largo, Maryland
  - John R. Graham Headache Center Brigham and Women's Faulkner Hospital, Boston, Massachusetts
  - BTC of New Bedford, New Bedford, Massachusetts
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Clinical Research Institute, Minneapolis, Minnesota
  - Synexus Usa, Bay Saint Louis, Mississippi
  - The Headache Center, Ridgeland, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC., Springfield, Missouri
  - Synexus Clinical Research US, Inc., Omaha, Nebraska
  - Nevada Headache Institute, Las Vegas, Nevada
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Dent Neurologic Institute, Amherst, New York
  - Northwell Health, Great Neck, New York
  - Montefiore Medical Center, The Bronx, New York
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - Guilford Neurologic Associates, Inc, Greensboro, North Carolina
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - Wilmington Health, PLLC, Wilmington, North Carolina
  - Piedmont Medical Research of Winston-Salem, Winston-Salem, North Carolina
  - Synexus Clinical Research US, Inc., Akron, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Patient Priority Clinical Sites, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Sentral Clinical Research Services, Cincinnati, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - Family Physicians Associates, Lyndhurst, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Centennial Health-Synexus, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, Tulsa, Oklahoma
  - Oregon Center for Clinical Investigations, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Preferred Primary Care Physicians, Jacob Murphy, Uniontown, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Partners in Clinical Research, Cumberland, Rhode Island
  - Ocean State Clinical Research Partners, Lincoln, Rhode Island
  - Primary Care Associates/Synexus Clinical, Anderson, South Carolina
  - Synexus Clinical Research US, Inc, Anderson, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Hillcrest Family Practice, Simpsonville, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - CNS Healthcare - Memphis, Memphis, Tennessee
  - Psychiatry & Psychotherapy Partners Austin, Austin, Texas
  - Tekton Research, Austin, Texas
  - Synexus-US, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Ventavia Research Group, Fort Worth, Texas
  - Centex Studies, Inc., Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Synexus Clinical Research US, Inc., San Antonio, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - Synexus-US, Murray, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - J. Lewis Research, Inc., South Jordan, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - National Clinical Research, Inc, Richmond, Virginia
  - Sentara Family Medicine Physicians, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource and Core Clinical Research, Everett, Washington
  - The Polyclinic, Seattle, Washington
  - Puget Sound Neurology, Tacoma, Washington

REFERENCES:
- [Derived] Goadsby PJ, Jurgens TP, Brand-Schieber E, Nagy K, Liu Y, Boinpally R, Stodtmann S, Trugman JM. Efficacy of ubrogepant and atogepant in males and females with migraine: A secondary analysis of randomized clinical trials. Cephalalgia. 2025 Feb;45(2):3331024251320610. doi: 10.1177/03331024251320610. PMID 39982105
- [Derived] Lipton RB, Gandhi P, Tassorelli C, Reuter U, Harriott AM, Holle-Lee D, Gottschalk CH, Neel B, Liu Y, Guo H, Stokes J, Nagy K, Dabruzzo B, Smith JH. Early Improvements With Atogepant for the Preventive Treatment of Migraine: Results From 3 Randomized Phase 3 Trials. Neurology. 2025 Jan 28;104(2):e210212. doi: 10.1212/WNL.0000000000210212. Epub 2024 Dec 23. PMID 39715475
- [Derived] Peterlin BL, Bond DS, Ailani J, Dodick DW, Liu Y, De Abreu Ferreira R, Smith JH, Dabruzzo B, Goadsby PJ, Trugman JM. Weight loss with atogepant during the preventive treatment of migraine: A pooled analysis. Cephalalgia. 2024 Dec;44(12):3331024241299753. doi: 10.1177/03331024241299753. PMID 39648629
- [Derived] Gottschalk C, Gandhi P, Pozo-Rosich P, Christie S, Tassorelli C, Stokes J, Liu Y, Luo L, Nagy K, Trugman JM, Lipton RB. Effect of preventive treatment with atogepant on quality of life, daily functioning, and headache impact across the spectrum of migraine: Findings from three double-blind, randomized, phase 3 trials. Cephalalgia. 2024 Dec;44(12):3331024241300305. doi: 10.1177/03331024241300305. PMID 39648617
- [Derived] Lipton RB, Nahas SJ, Pozo-Rosich P, Bilchik T, McAllister P, Finnegan M, Liu Y, Chalermpalanupap N, Dabruzzo B, Dodick DW. Sustained response to atogepant in episodic migraine: post hoc analyses of a 12-week randomized trial and a 52-week long-term safety trial. J Headache Pain. 2024 May 21;25(1):83. doi: 10.1186/s10194-024-01783-6. PMID 38773375
- [Derived] Rizzoli P, Marmura MJ, Robblee J, McVige J, Sacco S, Nahas SJ, Ailani J, De Abreu Ferreira R, Ma J, Smith JH, Dabruzzo B, Ashina M. Safety and tolerability of atogepant for the preventive treatment of migraine: a post hoc analysis of pooled data from four clinical trials. J Headache Pain. 2024 Mar 11;25(1):35. doi: 10.1186/s10194-024-01736-z. PMID 38462625
- [Derived] Lipton RB, Pozo-Rosich P, Blumenfeld AM, Li Y, Severt L, Stokes JT, Creutz L, Gandhi P, Dodick D. Effect of Atogepant for Preventive Migraine Treatment on Patient-Reported Outcomes in the Randomized, Double-blind, Phase 3 ADVANCE Trial. Neurology. 2023 Feb 21;100(8):e764-e777. doi: 10.1212/WNL.0000000000201568. Epub 2022 Nov 17. PMID 36396451
- [Derived] Lipton RB, Pozo-Rosich P, Blumenfeld AM, Dodick DW, McAllister P, Li Y, Lu K, Dabruzzo B, Miceli R, Severt L, Finnegan M, Trugman JM. Rates of Response to Atogepant for Migraine Prophylaxis Among Adults: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Jun 1;5(6):e2215499. doi: 10.1001/jamanetworkopen.2022.15499. PMID 35675076
- [Derived] Schwedt TJ, Lipton RB, Ailani J, Silberstein SD, Tassorelli C, Guo H, Lu K, Dabruzzo B, Miceli R, Severt L, Finnegan M, Trugman JM. Time course of efficacy of atogepant for the preventive treatment of migraine: Results from the randomized, double-blind ADVANCE trial. Cephalalgia. 2022 Jan;42(1):3-11. doi: 10.1177/03331024211042385. Epub 2021 Sep 14. PMID 34521260
- [Derived] Ailani J, Lipton RB, Goadsby PJ, Guo H, Miceli R, Severt L, Finnegan M, Trugman JM; ADVANCE Study Group. Atogepant for the Preventive Treatment of Migraine. N Engl J Med. 2021 Aug 19;385(8):695-706. doi: 10.1056/NEJMoa2035908. PMID 34407343
- [Derived] Boinpally R, McNamee B, Yao L, Butler M, McGeeney D, Borbridge L, Periclou A. A Single Supratherapeutic Dose of Atogepant Does Not Affect Cardiac Repolarization in Healthy Adults: Results From a Randomized, Single-Dose, Phase 1 Crossover Trial. Clin Pharmacol Drug Dev. 2021 Sep;10(9):1099-1107. doi: 10.1002/cpdd.940. Epub 2021 May 4. PMID 33942560
- [Derived] Min KC, Kraft WK, Bondiskey P, Colon-Gonzalez F, Liu W, Xu J, Panebianco D, Mixson L, Dockendorf MF, Matthews CZ, Boinpally R. Atogepant Is Not Associated With Clinically Meaningful Alanine Aminotransferase Elevations in Healthy Adults. Clin Transl Sci. 2021 Mar;14(2):599-605. doi: 10.1111/cts.12917. Epub 2020 Nov 24. PMID 33142014

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants diagnosed with episodic migraine were enrolled in one of 4 treatment arms: placebo, or atogepant 10 mg once daily (QD), 30 mg QD, 60 mg QD in Double-blind (DB) Treatment Period.
Period: DB Treatment Period (Up to Week 12)
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg
Started | 223 | 222 | 230 | 235
Treated: Safety Population (Safety Population included all participants who received at least 1 dose of study intervention.) | 222 | 221 | 228 | 231
Completed (Out of 805 participants who completed DB Treatment Period, 683 participants did not complete follow-up since they rolled into study 3101-309-002 (NCT03939312), 183 entered Follow-Up Period.) | 201 | 193 | 207 | 204
Not Completed | 22 | 29 | 23 | 31
Not completed — Adverse Event | 6 | 9 | 4 | 6
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 9 | 8 | 10
Not completed — Lost to Follow-up | 3 | 3 | 4 | 5
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 4 | 5 | 7 | 8
Not completed — Reason Not Specified | 0 | 2 | 0 | 1
Period: Follow-Up Period (Weeks 12 to 16)
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg
Started | 46 | 54 | 38 | 45
Completed | 41 | 49 | 32 | 36
Not Completed | 5 | 5 | 6 | 9
Not completed — Withdrawal by Subject | 5 | 3 | 4 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0 | 3
Not completed — Protocol Deviation | 0 | 1 | 1 | 0
Not completed — Reason Not Specified | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg | Total
Number analyzed (Participants) | 222 | 221 | 228 | 231 | 902
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (12.81) | 41.4 (12.05) | 42.1 (11.68) | 42.5 (12.41) | 41.6 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 200 | 204 | 199 | 801
  Male | 24 | 21 | 24 | 32 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 1 | 3
  Asian | 2 | 2 | 1 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 24 | 34 | 38 | 28 | 124
  White | 194 | 181 | 185 | 192 | 752
  More than one race | 2 | 3 | 3 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 23 | 21 | 19 | 14 | 77
  Non-Hispanic | 199 | 200 | 209 | 217 | 825
Monthly Migraine Days [Mean (Standard Deviation); unit: migraine days per month] — A migraine day was any calendar day on which the participant experienced a migraine headache qualified by duration or acute symptomatic medication use. The monthly (4-week) migraine days was defined as the total number of reported migraine days in diary divided by total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable Baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the Double-blind Treatment Period.
  migraine days per month
    number analyzed (Participants) | 214 | 214 | 223 | 222 | 873
    (all) | 7.5 (2.39) | 7.5 (2.46) | 7.9 (2.32) | 7.8 (2.31) | 7.6 (2.37)
Monthly Headache Days [Mean (Standard Deviation); unit: headache days per month] — A headache day is any calendar day on which the participant experienced a headache qualified by duration or acute symptomatic medication use. The monthly (4-week) headache days were defined as the total number of reported headache days in the diary divided by the total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable Baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the Double-blind Treatment Period.
  headache days per month
    number analyzed (Participants) | 214 | 214 | 223 | 222 | 873
    (all) | 8.4 (2.55) | 8.4 (2.75) | 8.8 (2.62) | 9.0 (2.56) | 8.7 (2.63)
Monthly Acute Medication Use [Mean (Standard Deviation); unit: acute medication use days per month] — The monthly (4-week) acute medication use days was defined as the total number of reported acute medication use days in the diary divided by the total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable Baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the Double-blind Treatment Period.
  acute medication use days per month
    number analyzed (Participants) | 214 | 214 | 223 | 222 | 873
    (all) | 6.5 (3.15) | 6.6 (2.99) | 6.7 (3.02) | 6.9 (3.17) | 6.7 (3.08)
MSQ v2.1 Role Function-Restrictive Domain Score [Mean (Standard Deviation); unit: score on a scale] — Migraine-Specific Quality of Life Questionnaire, Version 2.1 (MSQ v2.1) is 14-item questionnaire to measure health-related quality-of-life impairments attributed to migraine, divided in 3 domains: role function-restrictive: how migraines limit daily social and work-related activities; role function-preventive: how migraines prevent these activities; and emotional function domain: emotions associated with migraines, using a 6-point scale, 1=none of the time and 6=all of the time. Domain scores were rescaled from 0 to 100, with higher scores indicating better migraine specific quality of life. Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable Baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the Double-blind Treatment Period. Number analyzed is the number of participants available for the analyses at Baseline.
  score on a scale
    number analyzed (Participants) | 213 | 212 | 222 | 222 | 869
    (all) | 46.8 (19.67) | 44.9 (21.37) | 44.0 (19.61) | 46.8 (20.36) | 45.6 (20.26)
Daily Activities Domain Score of the Activity Impairment in Migraine- Diary (AIM-D) [Mean (Standard Deviation); unit: score on a scale] — AIM-D is a 9-item PRO measure that assesses the impact of migraine on performance of daily activities and physical impairment using a 6-point rating scale where 0=not difficult at all, 1=a little difficult, 2=somewhat difficult, 3=very difficult, 4=extremely difficult, and 5=I could not do it at all. The raw scores were transformed to 0-100 scale, with higher scores indicating greater impact of migraine. Baseline was defined as the monthly (averaged for a month) scores during the last 28 days. Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable Baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the Double-blind Treatment Period. Number analyzed is the number of participants available for the analyses at Baseline.
  score on a scale
    number analyzed (Participants) | 188 | 191 | 188 | 192 | 759
    (all) | 15.2 (8.25) | 15.5 (8.85) | 16.9 (8.02) | 15.9 (8.34) | 15.9 (8.38)
Monthly Physical Impairment Domain Score of the AIM-D [Mean (Standard Deviation); unit: score on a scale] — AIM-D is a 9-item PRO measure that assesses the impact of migraine on performance of daily activities and physical impairment using a 6-point rating scale where 0=not difficult at all, 1=a little difficult, 2=somewhat difficult, 3=very difficult, 4=extremely difficult, and 5=I could not do it at all. The raw scores were transformed to 0-100 scale, with higher scores indicating greater impact of migraine. Baseline was defined as the monthly (averaged for a month) scores during the last 28 days. Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable Baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the Double-blind Treatment Period. Number analyzed is the number of participants available for the analyses at Baseline.
  score on a scale
    number analyzed (Participants) | 188 | 191 | 188 | 192 | 759
    (all) | 11.2 (8.11) | 11.7 (8.46) | 13.0 (8.00) | 11.6 (7.85) | 11.9 (8.12)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Monthly Migraine Days Across the 12-Week Treatment Period
Description: Participants recorded daily duration of migraine in a diary. A migraine day was any calendar day on which the participant experienced a migraine headache qualified by duration or acute symptomatic medication use. The monthly (4-week) migraine days was defined as the total number of reported migraine days in diary divided by total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Baseline was defined as the number of migraine days during the last 28 days of the Baseline phase, from Day -28 to -1. Negative change from Baseline indicates improvement. A Mixed-effects model for repeated measures (MMRM) was used for analysis.
Time Frame: Baseline (Day -28 to Day -1) to Week 12
Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable Baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the Double-blind Treatment Period.
Measure: Least Squares Mean (Standard Error); unit: migraine days per month
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg
Number analyzed (Participants) | 214 | 214 | 223 | 222
migraine days per month | -2.48 (0.210) | -3.69 (0.210) | -3.86 (0.206) | -4.20 (0.206)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — MMRM model included Baseline monthly migraine days as a covariate, treatment group and visit (month) as fixed factors, and treatment group-by-visit and Baseline-by-visit as interaction terms, with an unstructured covariance matrix; Least Squares Mean Difference = -1.21, 95% CI 2-sided [-1.78 to -0.64], Standard Error of Mean 0.291
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.38, 95% CI 2-sided [-1.94 to -0.82], Standard Error of Mean 0.287
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.72, 95% CI 2-sided [-2.28 to -1.15], Standard Error of Mean 0.288

2. Secondary Outcome: Change From Baseline in Mean Monthly Headache Days Across the 12-Week Treatment Period
Description: Participants recorded daily total duration of a headache in a diary. A headache day is any calendar day on which the participant experienced a headache qualified by duration or acute symptomatic medication use. The monthly (4-week) headache days were defined as the total number of reported headache days in the diary divided by the total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Baseline was defined as the number of migraine days during the last 28 days of the Baseline phase, from Day -28 to -1. Negative change from Baseline indicates improvement. MMRM was used for analysis.
Time Frame: Baseline (Day-28 to Day -1) to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: headache days per month
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg
Number analyzed (Participants) | 214 | 214 | 223 | 222
headache days per month | -2.52 (0.225) | -3.94 (0.225) | -4.04 (0.221) | -4.23 (0.221)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.42, 95% CI 2-sided [-2.03 to -0.81], Standard Error of Mean 0.311
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.53, 95% CI 2-sided [-2.13 to -0.92], Standard Error of Mean 0.307
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.71, 95% CI 2-sided [-2.32 to -1.10], Standard Error of Mean 0.309

3. Secondary Outcome: Change From Baseline in Mean Monthly Acute Medication Use Days Across the 12-Week Treatment Period
Description: Participants recorded allowed medication(s) to treat an acute migraine in the daily diary. The monthly (4-week) acute medication use days was defined as the total number of reported acute medication use days in the diary divided by the total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Baseline was defined as the number of acute medication use days during the last 28 days of the Baseline phase, from Day -28 to -1. A negative change from Baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline (Day-28 to Day -1) to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: acute medication use days per month
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg
Number analyzed (Participants) | 214 | 214 | 223 | 222
acute medication use days per month | -2.35 (0.184) | -3.66 (0.183) | -3.68 (0.180) | -3.85 (0.180)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.31, 95% CI 2-sided [-1.81 to -0.82], Standard Error of Mean 0.254
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.33, 95% CI 2-sided [-1.82 to -0.83], Standard Error of Mean 0.251
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.50, 95% CI 2-sided [-2.00 to -1.01], Standard Error of Mean 0.252

4. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction (Improvement) in 3-month Average of Monthly Migraine Days
Description: Participants recorded daily duration of migraine in a diary. A migraine day was any calendar day on which the participant experienced a migraine headache qualified by duration or acute symptomatic medication use. The monthly (4-week) migraine days is equal to total number of reported migraine days in diary divided by total number of days with diary records in each 4-week period multiplied by 28. Each 4-week period was averaged.
Time Frame: Baseline (Day -28 to Day -1) to Week 12
Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable Baseline period (Day -28 to Day -1) of eDiary data, and had at least 1 evaluable post-baseline 4-week period (Weeks 1-4, 5-8, and 9-12) of eDiary data during the Double-blind Treatment Period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg
Number analyzed (Participants) | 214 | 214 | 223 | 222
percentage of participants | 29.0 | 55.6 | 58.7 | 60.8
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg; Test type: Superiority; p < .0001, Regression, Logistic — Odds ratio and p-value was based on logistic regression with treatment group, Baseline value, and prior exposure to a migraine prevention medications with proven efficacy as explanatory variables; Odds Ratio (OR) = 3.06, 95% CI 2-sided [2.05 to 4.56]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg; Test type: Superiority; p < .0001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 3.53, 95% CI 2-sided [2.37 to 5.26]
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < .0001, Regression, Logistic — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 3.82, 95% CI 2-sided [2.56 to 5.71]

5. Secondary Outcome: Change From Baseline in Migraine-Specific Quality of Life Questionnaire, Version 2.1 (MSQ v2.1) Role Function-Restrictive Domain Score at Week 12
Description: MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality-of-life impairments attributed to migraine in the past 4 weeks. It is divided into three domains: role function-restrictive (questions 1-7, score range 7 to 42) assesses how migraines limit one's daily social and work-related activities; role function-preventive (questions 8-11, score ranges 4 to 24) assesses how migraines prevent these activities; and the emotional function (questions 12-14, score ranges 3 to 18) domain assesses the emotions associated with migraines. Participants respond to items using a 6-point scale where 1=none of the time and 6=all of the time. Raw dimension scores are computed as a sum of item responses and rescaled to a 0 to 100 scale, where higher scores from Baseline indicate better quality of life. MMRM was used for the analysis.
Time Frame: Baseline (Day 1) to Week 12
Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable Baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period of eDiary data during the Double-blind Treatment Period. Overall number analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg
Number analyzed (Participants) | 198 | 186 | 203 | 201
score on a scale | 20.45 (1.617) | 30.35 (1.639) | 30.53 (1.593) | 31.25 (1.591)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 9.90, 95% CI 2-sided [5.45 to 14.36], Standard Error of Mean 2.270
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 10.08, 95% CI 2-sided [5.71 to 14.46], Standard Error of Mean 2.229
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 10.80, 95% CI 2-sided [6.42 to 15.18], Standard Error of Mean 2.231

6. Secondary Outcome: Change From Baseline in Mean Monthly Performance of Daily Activities Domain Score of the Activity Impairment in Migraine-Diary (AIM-D) Across the 12-Week Treatment Period
Description: The AIM-D is a 9-item PRO measure that assesses the impact of migraine on the performance of daily activities and physical impairment using a 6-point rating scale where 0=not difficult at all, 1=a little difficult, 2=somewhat difficult, 3=very difficult, 4=extremely difficult, and 5=I could not do it at all. The raw performance of daily activities domain scores were transformed to 0-100 scale, with higher scores indicating greater impact of migraine (higher disease burden). Baseline was defined as the monthly (averaged for a month) performance of daily activities domain score during the last 28 days of the Baseline period from Day -28 to -1. MMRM was used for the analysis.
Time Frame: Baseline (Day -28 to Day -1) to Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg
Number analyzed (Participants) | 178 | 182 | 181 | 178
score on a scale | -6.09 (0.504) | -7.28 (0.500) | -8.63 (0.502) | -9.41 (0.504)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg; Test type: Superiority; p = 0.0856, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.19, 95% CI 2-sided [-2.56 to 0.17], Standard Error of Mean 0.693
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg; Test type: Superiority; p = 0.0003, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -2.54, 95% CI 2-sided [-3.91 to -1.18], Standard Error of Mean 0.694
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -3.32, 95% CI 2-sided [-4.68 to -1.96], Standard Error of Mean 0.694

7. Secondary Outcome: Change From Baseline in Mean Monthly Physical Impairment Domain Score of the Activity Impairment in Migraine- Diary (AIM-D) Across the 12-Week Treatment Period
Description: The AIM-D is a 9-item PRO measure that assesses the impact of migraine on the performance of daily activities and physical impairment using a 6-point rating scale where 0=not difficult at all, 1=a little difficult, 2=somewhat difficult, 3=very difficult, 4=extremely difficult, and 5=I could not do it at all. The raw physical impairment domain scores were transformed to 0-100 scale, with higher scores indicating greater impact of migraine (higher disease burden). Baseline was defined as the monthly (averaged for a month) physical impairment domain score during the last 28 days of the Baseline period from Day -28 to -1. MMRM was used for the analysis.
Time Frame: Baseline (Day -28 to Day -1) to Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg
Number analyzed (Participants) | 178 | 182 | 181 | 178
score on a scale | -4.03 (0.439) | -5.11 (0.436) | -6.02 (0.438) | -6.49 (0.439)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 10 mg; Test type: Superiority; p = 0.0743, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.08, 95% CI 2-sided [-2.27 to 0.11], Standard Error of Mean 0.605
Statistical Analysis 2: Comparison: Placebo vs Atogepant 30 mg; Test type: Superiority; p = 0.0011, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.99, 95% CI 2-sided [-3.18 to -0.80], Standard Error of Mean 0.606
Statistical Analysis 3: Comparison: Placebo vs Atogepant 60 mg; Test type: Superiority; p < .0001, Mixed-effects Model for Repeated Measure — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -2.46, 95% CI 2-sided [-3.65 to -1.28], Standard Error of Mean 0.605

ADVERSE EVENTS:
Time Frame: From first dose of study drug through end of study (Up to 16 weeks)
Description: All-Cause Mortality is reported for all randomized participants. Safety Population, all participants who received at least 1 dose of study intervention, was used to determine the number of participants at risk for Serious Adverse Events and Other Adverse Events.
Arm/Group | Placebo | Atogepant 10 mg | Atogepant 30 mg | Atogepant 60 mg
All-Cause Mortality (participants affected / at risk) | 0/223 | 0/222 | 0/230 | 0/235
Serious Adverse Events (participants affected / at risk) | 2/222 | 2/221 | 0/228 | 0/231
Other Adverse Events (participants affected / at risk) | 15/222 | 34/221 | 37/228 | 32/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=222) | Atogepant 10 mg (N=221) | Atogepant 30 mg (N=228) | Atogepant 60 mg (N=231)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Negative pressure pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=222) | Atogepant 10 mg (N=221) | Atogepant 30 mg (N=228) | Atogepant 60 mg (N=231)
Constipation (Gastrointestinal disorders) | 1 | 17 | 16 | 16
Nausea (Gastrointestinal disorders) | 4 | 11 | 10 | 14
Upper respiratory tract infection (Infections and infestations) | 10 | 9 | 13 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-05-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT03777059/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT03777059/SAP_001.pdf